CLINICAL TRIAL: NCT05106218
Title: Assessment of the SurroundScope in Urologic Surgical Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: 270Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL 466
Record Dates: First submitted 2021-10-07; First posted 2021-11-03 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-11

CONDITIONS: Partial Nephrectomy; Nephrectomy; Laparoscopy

STUDY DESIGN:
Intervention Model Description: For laparoscopic camera system to be used in urological surgeries, the SurroundScope, 270-degree angle videoscope (270Surgical, Israel) is used. This will be compared to the standard laparoscopic system use.
  The study will evaluate standard urological surgeries using the 270Surgical system vs same procedures using the standard scope. The procedure will be performed according to the institution's standard of care, using the SurroundScope or the standard scope for visualization. Each surgery will be captured on video.
Who Masked: Participant
Masking Description: Patients are not aware of the laparoscopic system that will be used during the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SurroundScope (Experimental): For laparoscopic camera system, the SurroundScope, 270-degree angle videoscope (270Surgical, Israel) is used
  Interventions: Device: SurroundScope
- Standard laparoscope (Active Comparator): For laparoscopic camera system, the Standard laparoscope that is in a standard use at the medical center is used
  Interventions: Device: Standard Laparoscope

INTERVENTIONS:
Device: SurroundScope — The procedure will be performed according to the institution's standard of care, using the SurroundScope for visualization.
  Other Names: 270System
  Arms: SurroundScope
Device: Standard Laparoscope — The procedure will be performed according to the institution's standard of care, using the Standard laparoscope for visualization.
  Arms: Standard laparoscope

SUMMARY:
The aim of this study is to evaluate standard urological surgeries using the 270Surgical system vs same procedures using the standard scope

DETAILED DESCRIPTION:
The tremendous popularity of the laparoscopic surgeries is balanced with its tradeoffs - the needs for an excellent intracavitary visualization along with a surgeon skill set capable of performing these, often more technically challenging procedures. Image quality has improved, but there are still various restrictions to images captured by the lens at the tip of a long tubular laparoscope. 270Surgical developed a 270 degree angle scope to overcome these unmet needs and improve the image quantity and extent during laparoscopy. The study will compare the use of the 270Surgical system (The "SurroundScope") to standard laparoscope during partial nephrectomy and nephrectomy urological surgeries;

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Capable of giving informed consent.
* Scheduled for laparoscopic urologic surgery: Partial nephrectomy, Nephrectomy

Exclusion Criteria:

* Unfit for surgery: concomitant disorders incompatible with the study or surgery (at the discretion of the investigator)
* Patients with contraindications to undergo laparoscopic surgery.
* Patients with American Society of Anesthesiology (ASA) class* >3
* Advanced cirrhosis with failure of hepatic function
* Patients who have participated in another interventional clinical study in the last month.
* Pregnancy
* Unable to consent (due to cultural, language or neurological barriers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Analysis of the efficient work time with the standard scope and the SurroundScope - Time of surgery | During the surgery - Since the first incision performed till the last incision is closed
  Data collected include - skin to skin time of surgery
Analysis of the efficient work time with the standard scope and the SurroundScope - tools and ports Visibility time | During the surgery - Since the first incision performed till the last incision is closed
  Data collected include - Visibility time of tools and ports in the Field of view
Analysis of the efficient work time with the standard scope and the SurroundScope - time of scope removals | During the surgery - Since the first incision performed till the last incision is closed
  Data collected include - Time of scope removals during the case to clear smoke or fog

SECONDARY OUTCOMES:
Time of defined surgical tasks - port placement time | During the defined surgical task
  Time to complete port placement will be measured
Time of defined surgical tasks - transection time | During the defined surgical task
  Time to transection of renal artery & Vein with stapler will be measured
Time of defined surgical tasks - clamp time | During the defined surgical task
  Clamp time during partial nephrectomy will be measured

OTHER OUTCOMES:
Adverse events | During the surgery - Since the first incision performed till the last incision is closed
  Amount of intraoperative adverse event
Length of stay | Since the surgery completion to discharge from the medical center
  Length of stay at the hospital following the surgery in days
Surgeon's perception 270surgical | Immediately following the surgery is completed
  Surgeon's perception of the 270surgical System - Assessed by a multi-question subjective questionnaire completed in the OR, immediately after the case, by the surgeon and the camera person and constructed on a Likert-type, 5-point scale (1=Strongly disagree, 2=Disagree, 3=Neither agree or disagree, 4=Agree, 5=Strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Nado, MD, Principal Investigator — Rabin Medical Center, 39 Jabotinski St., Petah Tikva 49100
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No